CLINICAL TRIAL: NCT03705429
Title: A Multi-Centre Randomized Study Comparing Two Standard of Care Adjuvant Chemotherapy Regimens for Lower Risk HER-2 Positive Breast Cancer
Brief Title: A Study Comparing Two Standard of Care Adjuvant Chemotherapy Regimens for Lower Risk HER-2 Positive Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: The Ottawa Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REaCT-Low Risk HER-2
Record Dates: First submitted 2018-09-24; First posted 2018-10-15 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Cyclophosphamide; Trastuzumab; Paclitaxel

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TC-H Chemotherapy (Active Comparator): Docetaxel 75 mg/m2, Cyclophosphamide 600 mg/m2 and Trastuzumab 8 mg/kg followed by 6 mg/kg Day 1 every 21 days for 4 cycles. Trastuzumab 6 mg/kg Day 1 every 21 days to complete 1 year of Trastuzumab therapy.
  Interventions: Drug: TC-H x Paclitaxel (P) + Trastuzumab(T)
- Paclitaxel(P) + Trastuzumab(T) (Placebo Comparator): Paclitaxel 80 mg/m2 weekly for 12 weeks and Trastuzumab 8 mg/kg followed by 6 mg/kg Day 1 every 21 days for 4 cycles. Trastuzumab 6 mg/kg Day 1 every 21 days to complete 1 year of Trastuzumab therapy. Alternatively Trastuzumab 4 mg/kg followed by 2 mg/kg weekly to complete 1 year of treatment can be used.
  Interventions: Drug: TC-H x Paclitaxel (P) + Trastuzumab(T)

INTERVENTIONS:
Drug: TC-H x Paclitaxel (P) + Trastuzumab(T) — chemotherapy
  Other Names: Docetaxel, Cyclophosphamide and Trastuzumab; Paclitaxel and Trastuzumab

SUMMARY:
Multi-center, open-label, randomized trial of patients with low-risk, HER2+ disease, who will receive adjuvant taxane-based chemotherapy (i.e. docetaxel and cyclophosphamide with trastuzumab [TC-H] or weekly paclitaxel with trastuzumab [P-H]) at the standard approved doses, aiming to gather more information regarding cost-effectiveness, toxicity, quality of life (QoL), patient reported outcomes and clinical benefits of the two treatment strategies.

DETAILED DESCRIPTION:
Multi-center, open-label, randomized trial of patients with low-risk, HER2+ disease, who will receive adjuvant taxane-based chemotherapy (i.e. docetaxel and cyclophosphamide with trastuzumab [TC-H] or weekly paclitaxel with trastuzumab [P-H]) at the standard approved doses. The primary objective is to estimate the feasibility of opening a pragmatic clinical trial with an Integrated Consent Model Secondary objectives are: Compare adverse events/ toxicity profile between the two different approaches (i.e. neutropenia, peripheral neuropathy, treatment-related hospitalizations, proportion of patients completing the chemotherapy component of their treatment); Estimate the cost of each chemotherapy regimen and potential cost-effectiveness analysis from the perspective of Canada's health care system; Evaluate the impact on activities of daily living as reflected by self-reported fatigue and pain using the FACT-Taxane and FACIT-Fatigue scores. In this study, the investigator will obtain oral consent using the prepared REB approved Consent Script. If the patient agrees to participate, the physician will dictate in the progress note they have had the above conversation with the patient. There will be no need for the patient to sign an informed consent form.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HER-2 positive early stage breast cancer for whom TC-H or weekly P-H is being considered.
* Able to provide verbal consent.
* Willing to complete study related-questionnaires

Exclusion Criteria:

* Unable to give informed consent or complete questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-05-11 (Actual)

PRIMARY OUTCOMES:
Feasibility of performing a pragmatic clinical trial with an Integrated Consent Model. | up to 12 months.
  Feasibility of performing this study will be measured with 2 composite endpoints: number of patients who received either TC-H or P-H chemotherapy compared to the number of participants who were approached to enter the study.

SECONDARY OUTCOMES:
Adverse events/ toxicity profile between the two different approaches. | up to 12 months.
  Toxicity profile (NCI CTC version 4.1)
Cost of each chemotherapy regimen and potential cost-effectiveness analysis. | up to 12 months.
  Health system cost of each chemotherapy regimen.
Cost-effectiveness analysis. | up to 12 months.
  Cost per one quality-adjusted life year (QALY) gained.
Cost-effectiveness analysis. | up to 12 months.
  Use of primary or secondary febrile neutropenia prophylaxis.
Quality of life as reflected by self-reported fatigue using FACIT-Fatigue scores. | up to 12 months.
  Functional Assessment of Chronic Illness Therapy -Fatigue (FACIT-Fatigue) scores
Quality of life as reflected by self-reported pain using FACT-Taxane scores | up to 12 motnhs.
  Functional Assessment of Cancer Therapy-Taxane Scores.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Fernandes, M.D., Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (3):
- Canada (3):
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario

IPD SHARING:
Plan to Share IPD: No